CLINICAL TRIAL: NCT06786208
Title: Real-world Study of Sunvozertinib Treatment in Locally Advanced or Metastatic EGFR-Mutant NSCLC After EGFR-TKI Treatment Failure
Brief Title: Real-world Study of Sunvozertinib Treatment in Advanced EGFR-Mutant NSCLC After EGFR-TKI Treatment Failure
Status: Not yet recruiting | Type: Observational
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2024-388; 2024-388 (Other: Henan cancer hospital affiliated cancer hospital of zhengzhou university)
Record Dates: First submitted 2025-01-15; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-11

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non Small Cell Lung Cancer; Sunvozertinib; EGFR
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- sunvozertinib treatment cohort: Patients: locally advanced or metastatic NSCLC with EGFR-sensitive mutations who have been previously treated with EGFR-TKIs and PD for last therapy.
  Investigators will assess patients whether to be suitable for sunvozertinib treatment. And this study will evaluate the safety and efficacy.
  Interventions: Drug: Sunvozertinib

INTERVENTIONS:
Drug: Sunvozertinib — sunvozertinb, a EGFR-TKI, 300mg QD oral

SUMMARY:
Observe the efficacy and safety of sunvozertinib in the real world in the treatment of EGFRm aNSCLC patients with previous EGFR-TKI treatment

DETAILED DESCRIPTION:
Locally advanced or metastatic NSCLC with EGFR-sensitive mutations who have been previously treated with EGFR-TKIs and PD for last therapy can be involved in this study. Investigators will assess patients whether to be suitable for sunvozertinib treatment. And this study will evaluate the safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. To provide a signed and dated, written informed consent.
2. Age ≥ 18 years old
3. Histologically or cytologically confirmed non-squamous NSCLC with documented EGFR mutations from a local laboratory
4. EGFR-sensitive mutations including exon 19 deletion and exon 21 L858R mutated，at least one line chemotherapy and progress again
5. Predicted life expectancy ≥ 12 weeks
6. Adequate organ system function:
7. Patient must have measurable disease according to RECIST 1.1. -

Exclusion Criteria:

1. Spinal cord compression or meningeal metastasis
2. Not Recover from AEs caused by previous treatment yet
3. A history of stroke or intracranial hemorrhage within 6 months prior to initial dosing.
4. Any severe or poorly controlled systemic disease per investigator's judgment .active infections, including but not limited to hepatitis B (HBV), hepatitis C HCV, and human immunodeficiency HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Locally advanced or metastatic NSCLC with EGFR-sensitive mutations who have been previously treated with EGFR-TKIs and PD for last therapy can be involved in this study. Investigators will assess patients whether to be suitable for sunvozertinib treatment.
Sampling Method: Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Time from first dose to last dose, up to 24 month
  assess the proportion of subjects who have a complete response (CR) or a partial response (PR)]

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Time from first dose to first documented disease progression assessed by investigator or death due to any cause up to 24 month
  To assess anti-tumor activity of Sunvozertinib according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by investigator
Overall survival (OS) | Time Frame: Time from first dose to the death of the subject due to any cause assessed up to 36 months.
  To assess anti-tumor activity of Sunvozertinib according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by investigator

CONTACTS AND LOCATIONS:
Locations (1):
- Qiming Wang, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No